CLINICAL TRIAL: NCT00106743
Title: Natural History and Genetic Studies of Usher Syndrome
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050096; 05-EI-0096
Record Dates: First submitted 2005-03-29; First posted 2005-03-30 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-04-30

CONDITIONS: Retinitis Pigmentosa Syndromic; Congenital Deafness; Usher Syndrome; Retinitis Pigmentosa and Deafness; Retinitis Pigmentosa
Keywords: Usher Syndrome; Retinitis Pigmentosa; Congenital Deafness
MeSH Terms: conditions — Usher Syndromes; Retinitis Pigmentosa; Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will explore clinical and genetic aspects of Usher syndrome, an inherited disease causing deafness or impaired hearing, visual problems, and, in some cases, unsteadiness or balance problems. Patients with type 1 Usher syndrome usually are deaf from birth and have speech and balance problems. Patients with type 2 disease generally are hearing impaired but have no balance problems. Patients with type 3 disease have progressive hearing loss and balance problems. All patients develop retinitis pigmentosa, an eye disease that causes poor night vision and eventually, blindness.

Patients of any age with Usher syndrome may be eligible for this study. Patients who have had eye and hearing evaluations are asked to send their medical records to the research team at the National Eye Institute (NEI) for review. They are also asked to have a blood sample drawn by a medical professional and sent to NEI for genetic analysis. Finally, they are interviewed about their family histories, particularly about other relative with eye disease. Patients who have not been evaluated previously have the following tests and procedures at NIH:

* Family medical history, especially regarding eye disease. A family tree is drawn.
* Blood draw for genetic studies of Usher syndrome.
* Eye examination to assess visual acuity and eye pressure, and to examine pupils, lens, retina, and eye movements.
* Electroretinogram (ERG) to test the function of visual cells. Wearing eye patches, the patient sits in a dark room for 30 minutes. Electrodes are taped to the forehead and the eye patches are removed. The surface of the eye is numbed with eye drops and contact lenses are placed on the eyes. The patient looks inside a hollow, dark globe and sees a series of light flashes. Then a light is turned on inside the globe and more flashes appear. The contact lenses sense small electrical signals generated by the retina when the light flashes.
* Fluorescein angiography to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Hearing tests to help determine the patient's type of Usher syndrome. Tests to evaluate hearing include examination of both ears with an otoscope, evaluation of the middle ear and inner ear, and hearing tests using earphones that deliver tones and words the subject listens and responds to.
* Vestibular testing for balance function. Balance testing involves three procedures:

Videonystagmography: This test records eye movements with little cameras. First the patient follows the movements of some small lights. Next, while wearing goggles, the patient lies on an exam table and turns to the right and left. Lastly, a soft stream of air is blown into the patient's ears four times, once in each ear with cool air and once in each ear with warm air.

Rotary chair test: With electrodes placed on the forehead, the patient sits in a rotary chair in a dark room. Several red lights appear on the wall of the room and the patient follows the lights as they move back and forth. Then the chair turns at several speeds, all slower than a merry-go-round.

Vestibular evoked potential: Electrodes are placed behind the patient's ear and at the base of the neck. Seated in a reclining chair and wearing earphones, the patient hears a brief series of loud clicking sounds. When the sounds are on, the patient is asked to lift his or her head up a few inches from the chair. The electrodes record information from the muscles in the neck as the sounds enter the ear.

DETAILED DESCRIPTION:
Background and objectives:

The Usher syndromes are a group of clinically variable and genetically heterogeneous autosomal recessive syndromes. On the basis of clinical findings, at least three types exist. Patients with Usher type I are born deaf, have vestibular problems, and are thought to perceive night blindness in early childhood. Patients with Usher type II are born with a hearing deficit but are able to develop intelligible speech, do not have balance problems; night vision problems, and visual field changes are noted later. Patients with Usher type III are born with relatively good hearing that deteriorates over a decade or more; they can have progressive balance problems and they report night blindness in childhood or teens. Seven genes have been mapped so far for Usher type I while five of these genes have been identified. For Usher type II, four genes have been mapped and three of these have been identified while there is one cloned gene for Usher type III. Quite a lot of information is still unknown regarding the genetic nature of this syndrome. The picture of the three clinical types of Usher syndrome has also not been well studied up to this point and cross sectional studies seems to be the only source of the information available so far, regarding the natural history of the disease. The aim of this protocol is to better study the natural history of the disease and also make specific genotype-phenotype correlations.

Study population:

A total of 200 participants, including patients affected with all three clinical types of Usher syndrome and up to 200 unaffected relatives will be enrolled to the protocol. Unaffected family members, primarily parents and siblings will be enrolled to provide a blood sample when considered helpful for linkage analysis. Family members will be considered unaffected if they have had a previous normal examination and they don t have any symptoms of decreased night or peripheral vision.

Methods:

Participants will undergo ophthalmologic, audiologic and vestibular evaluation in order to be clinically characterized. Blood will be obtained by all participating subjects for the molecular studies. Patients who cannot come to NIH or a collaborating Institution for participation will be asked to provide a blood sample for genotyping and a copy of their ophthalmologic, audiology and vestibular records, to classify phenotype. Each off-site participant will be consented over the phone by an NEI investigator. All participants will be requested to fill out a questionnaire.

Outcome measures:

Affected participants will be phenotypically categorized in one of the three clinical types based on audiology and vestibular findings

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible participants must:

1. have documented neurosensory hearing loss and retinitis pigmentosa and fulfill the clinical characteristics for USH1, USH2 and USH3 as defined by the Usher syndrome consortium. ; OR
2. be unaffected family members of a proband with Usher s syndrome, primarily parents and siblings. Family members will be considered unaffected by history if they have had previous normal ophthalmologic and hearing examinations and if they don't have decreased night or peripheral vision.

EXCLUSION CRITERIA:

Patients will be ineligible if they:

1. had an intrauterine infection, perinatal/congenital infections, or intrauterine and birth complications. These conditions can result in damage to both the auditory or visual system.
2. have concurrent inherited or acquired conditions that affect the visual and/or auditory system and significantly alter the phenotype.

Both affected and unaffected individuals will be ineligible if they:

1. Are unwilling or unable to provide a blood sample or unable to undergo the study procedures.
2. Are younger than 2 years old.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2005-03-21; Study Completion 2019-04-30

PRIMARY OUTCOMES:
The primary outcomes of interest are the probands genotype and phenotype. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wadih Zein, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Queens College of the City University of New York, New York, New York

REFERENCES:
- [Background] Smith RJ, Berlin CI, Hejtmancik JF, Keats BJ, Kimberling WJ, Lewis RA, Moller CG, Pelias MZ, Tranebjaerg L. Clinical diagnosis of the Usher syndromes. Usher Syndrome Consortium. Am J Med Genet. 1994 Mar 1;50(1):32-8. doi: 10.1002/ajmg.1320500107. PMID 8160750
- [Background] Keats BJ, Corey DP. The usher syndromes. Am J Med Genet. 1999 Sep 24;89(3):158-66. PMID 10704190
- [Background] Fishman GA, Kumar A, Joseph ME, Torok N, Anderson RJ. Usher's syndrome. Ophthalmic and neuro-otologic findings suggesting genetic heterogeneity. Arch Ophthalmol. 1983 Sep;101(9):1367-74. doi: 10.1001/archopht.1983.01040020369005. PMID 6604514